CLINICAL TRIAL: NCT04728464
Title: Evaluation of the Levels of Pain and Discomfort of 'Periodontally Accelerated Osteogenic Orthodontics' (PAOO) in the Leveling and Alignment of Crowded Lower Anterior Teeth: A Prospective Non-controlled Cohort Study
Brief Title: Pain, Acceptance, and Discomfort With Periodontally Accelerated Osteogenic Orthodontics (PAOO)
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-Ortho-01-2021
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Crowding of Anterior Mandibular Teeth
Keywords: Visual Analog Scale; Acceleration; moderate crowding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Periodontally Accelerated Osteogenic Orthodontics (PAOO): Patients will be treated by Periodontally Accelerated Osteogenic Orthodontics using fixed appliances.
  Interventions: Procedure: Periodontally Accelerated Osteogenic Orthodontics (PAOO)

INTERVENTIONS:
Procedure: Periodontally Accelerated Osteogenic Orthodontics (PAOO) — Fixed appliance will be placed for every patient, then surgical procedure will be applied after reflecting a full-thickness labial flap.

SUMMARY:
Patients will be examined in the Orthodontic Department of the University of Damascus Dental School. Patients who will be treated in conjunction with the PAOO procedure and subjects who will meet the inclusion criteria will be included then the initial diagnostic records (diagnostic gypsum models, internal and external oral photographs, as well as radiographic images) will be studied to ensure that the selection criteria will be accurately matched. This study aims to assess patients' acceptance of the PAOO procedure as well as the levels of pain and discomfort associated with this treatment.

DETAILED DESCRIPTION:
Surgical procedure associated with PAOO The surgery will be performed under local anesthesia and then full-thickness flaps will be reflected labially only from the distal surface of the lower right canine to the distal surface of the lower left canine, after washing the exposed alveolar bone with saline, then a selective cortical cutting will be performed using a piezosurgery and then the Bone-D® xenograft (particle size of 0.2 mm-1.0 mm) from Medpark (Busan, Korea) will be placed, then the wound will be sutured. Then a schedule will be set up to review the patient after 1, 7, 14, and 28 days to fill out questionnaires related to pain, acceptance, discomfort, satisfaction, and follow-up to orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Class I malocclusion with moderate crowding (4-6 mm of a tooth-size-arch-length-discrepancy).
2. Good oral hygiene and periodontal health.
3. No severe skeletal discrepancy.
4. Normal proclination for the upper and lower incisors.
5. No congenitally missing or extracted teeth (except for the third molars).

Exclusion Criteria:

1. Bimaxillary dentoalveolar severe protrusion.
2. Previous orthodontic treatment.
3. Subject with psychological abnormalities.
4. Subject with systemic diseases.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with malocclusion
  1. Crowding on the lower arch with a moderate degree (i.e., between 4 to six millimeters of a tooth-size-arch-length discrepancy).
  2. Class I malocclusion
  3. With no severe skeletal discrepancy.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in perception of pain | (1) one day following the beginning of the treatment, (2) after a week of the beginning of treatment, (3) after 2 weeks, (4) after 4 weeks
  Patients will be asked about their pain perception (item 1 of the first questionnaire).
  "How much pain did you have?" A standardized questionnaire to assess pain, acceptance, and discomfort during the first month of treatment based on a set of questions that will be answered by the Visual Analog Scale (VAS).
  The patient will specify a point on the line that expresses his feels, the score is determined by measuring the distance from the beginning until the point identified by the patient. The analog scale is a 100 mm horizontal line with two focal points at its beginning and end (0: there is no pain - 100: the worst pain).
Change in perception of discomfort | (1) one day following the beginning of the treatment, (2) after a week of the beginning of treatment, (3) after 2 weeks, (4) after 4 weeks
  Patients will be asked about their discomfort (item 2 of the first questionnaire).
  "How much discomfort did you have?" A standardized questionnaire to assess pain, acceptance, and discomfort during the first month of treatment based on a set of questions that will be answered by the Visual Analog Scale (VAS).
  The patient will specify a point on the line that expresses his feels, the score is determined by measuring the distance from the beginning until the point identified by the patient. The analog scale is a 100 mm horizontal line with two focal points at its beginning and end (0: there is no discomfort - 100: the worst discomfort).
Change in the feeling of swelling | (1) one day following the beginning of the treatment, (2) after a week of the beginning of treatment, (3) after 2 weeks, (4) after 4 weeks
  Patients will be asked about how much they feel swollen (item 3 of the first questionnaire).
  "How much swelling did you feel?" A standardized questionnaire to assess pain, acceptance, and discomfort during the first month of treatment based on a set of questions that will be answered by the Visual Analog Scale (VAS).
  The patient will specify a point on the line that expresses his feels, the score is determined by measuring the distance from the beginning until the point identified by the patient. The analog scale is a 100 mm horizontal line with two focal points at its beginning and end (0: there is no swelling - 100: the worst swelling).
Change in the difficulty of mastication | (1) one day following the beginning of the treatment, (2) after a week of the beginning of treatment, (3) after 2 weeks, (4) after 4 weeks
  Patients will be asked about the difficulty of mastication (item 4 of the first questionnaire).
  "How many difficulties in mastication did you have?" A standardized questionnaire to assess pain, acceptance, and discomfort during the first month of treatment based on a set of questions that will be answered by the Visual Analog Scale (VAS).
  The patient will specify a point on the line that expresses his feels, the score is determined by measuring the distance from the beginning until the point identified by the patient. The analog scale is a 100 mm horizontal line with two focal points at its beginning and end (0: there is no difficulty of mastication - 100: the worst difficulty of mastication).
Change in difficulty swallowing | (1) one day following the beginning of the treatment, (2) after a week of the beginning of treatment, (3) after 2 weeks, (4) after 4 weeks]
  Patients will be asked about how difficult it is to swallow (item 5 of the first questionnaire).
  "How many difficulties in swallowing did you feel?" A standardized questionnaire to assess pain, acceptance, and discomfort during the first month of treatment based on a set of questions that will be answered by the Visual Analog Scale (VAS).
  The patient will specify a point on the line that expresses his feels, the score is determined by measuring the distance from the beginning until the point identified by the patient. The analog scale is a 100 mm horizontal line with two focal points at its beginning and end (0: there is no difficulty swallowing - 100: the worst difficulty swallowing).
Change in the limits of opening the mouth | (1) one day following the beginning of the treatment, (2) after a week of the beginning of treatment, (3) after 2 weeks, (4) after 4 weeks
  Patients will be asked about the limits of the mouth opening limits (item 6 of the first questionnaire).
  "How much mouth limitation did you feel?" A standardized questionnaire to assess pain, acceptance, and discomfort during the first month of treatment based on a set of questions that will be answered by the Visual Analog Scale (VAS).
  The patient will specify a point on the line that expresses his feels, the score is determined by measuring the distance from the beginning until the point identified by the patient. The analog scale is a 100 mm horizontal line with two focal points at its beginning and end (0: there is no limitation in opening the mouth - 100: the worst limits in opening the mouth).
Change in the level of satisfaction with accelerated treatment | (1) after 4 weeks following the beginning of the treatment
  Patients will be asked about satisfaction with accelerated treatment (item 1 of the second questionnaire).
  "How much are you satisfied with your accelerated treatment?" A standardized questionnaire to assess pain, acceptance, and discomfort during the first month of treatment based on a set of questions that will be answered by the Visual Analog Scale (VAS).
  The patient will specify a point on the line that expresses his feels, the score is determined by measuring the distance from the beginning until the point identified by the patient. The analog scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no satisfaction with accelerated treatment - 100: best satisfaction with accelerated treatment).
Recommendation for the procedure | (1) after 4 weeks following the beginning of the treatment
  Patients will be asked about a friend's recommendation for this procedure (item 2 of the second questionnaire).
  "Would you recommend this procedure to a friend?" A standardized questionnaire to assess pain, acceptance, and discomfort during the first month of treatment based on a set of questions that will be answered. The scale is two-point (yes, no) and the patient will select one answer yes or no.
Taking any type of pain killers | (1) after 4 weeks following the beginning of the treatment
  Patients will be asked about taking any type of pain killers (item 3 of the second questionnaire).
  "Did you take any type of pain killers during the treatment?" A standardized questionnaire to assess pain, acceptance, and discomfort during the first month of treatment based on a set of questions that will be answered. The scale is two-point (Yes, No) and the patient will select one answer yes or no.
  If the patient's answer is (Yes), he is asked to specify the number of pain killers that he took during the treatment "when did you take pain killers? How many tablets as a whole?"

CONTACTS AND LOCATIONS:
Overall Officials: Hallaj I Alsino, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental; Mohammad Y Hajeer, DDS,MSc,PhD, Study Chair — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Issam Khoury, DDS,MSc,PhD, Study Director — Professor of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhattacharya P, Bhattacharya H, Anjum A, Bhandari R, Agarwal DK, Gupta A, Ansar J. Assessment of Corticotomy Facilitated Tooth Movement and Changes in Alveolar Bone Thickness - A CT Scan Study. J Clin Diagn Res. 2014 Oct;8(10):ZC26-30. doi: 10.7860/JCDR/2014/9448.4954. Epub 2014 Oct 20. PMID 25478442
- [Background] Chandra RV, Rachala MR, Madhavi K, Kambalyal P, Reddy AA, Ali MH. Periodontally accelerated osteogenic orthodontics combined with recombinant human bone morphogenetic protein-2: An outcome assessment. J Indian Soc Periodontol. 2019 May-Jun;23(3):257-263. doi: 10.4103/jisp.jisp_612_18. PMID 31143007
- [Background] Shoreibah EA, Ibrahim SA, Attia MS, Diab MM. Clinical and radiographic evaluation of bone grafting in corticotomy-facilitated orthodontics in adults. J Int Acad Periodontol. 2012 Oct;14(4):105-13. PMID 23210199
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984
- [Background] Wilcko WM, Wilcko T, Bouquot JE, Ferguson DJ. Rapid orthodontics with alveolar reshaping: two case reports of decrowding. Int J Periodontics Restorative Dent. 2001 Feb;21(1):9-19. PMID 11829041